CLINICAL TRIAL: NCT00049257
Title: A Phase II Trial of Paclitaxel and Carboplatin in the Treatment of Hormone-Refractory Prostate Cancer (HRPC)
Brief Title: Paclitaxel and Carboplatin in Treating Patients With Metastatic Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000258050; UCLA-0202092; BMS-UCLA-020209201; NCI-G02-2121
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Results first posted 2012-03-15 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2012-08

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Please see intervention descriptions
  Interventions: Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin — Administered Day 1 of each cycle. AUC=6.
  Other Names: Paraplatin
Drug: paclitaxel — administered Days 1, 8, and 15 of each cycle. 100mg/m2
  Other Names: Taxol

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining paclitaxel with carboplatin in treating patients who have metastatic prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the prostate-specific antigen (PSA) response rate and time to PSA progression in patients with metastatic hormone-refractory prostate cancer treated with paclitaxel and carboplatin.
* Determine the objective response rate, time to measurable or evaluable disease progression, and overall survival in patients treated with this regimen.
* Determine the safety and toxicity of this regimen in these patients.

OUTLINE: This is an open-label study.

Patients receive paclitaxel IV on days 1, 8, and 15 and carboplatin IV on day 1. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 4 weeks for 12 weeks and then every 2 months thereafter.

PROJECTED ACCRUAL: Approximately 60 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be informed of investigational nature of the study and written informed consent must be obtained prior to study entry
* Patients >18 years of age
* Patients with a histologic diagnosis of adenocarcinoma of the prostate
* Patients must have metastatic disease with progression despite androgen ablation. Patients who have not undergone orchiectomy must continue LHRH analogues. For patients receiving LHRH analogues their testosterone level must be < 50ng/dL
* Patients with bidimensionally measurable disease or bone metastases that is not progressive but who have a rising PSA are eligible
* Patients with an ECOG performance status <2
* Patients must have discontinued flutamide or nilutamide at least 4 weeks prior to the first day of treatment with evidence of progressive disease. Patients must have discontinued bicalutamide at least 6 weeks prior to registration with evidence of progressive disease
* Patients with adequate hematological, renal, and hepatic function as defined by the following required laboratory values:

  * While blood cell count: > 3,000/mm3
  * Absolute granulocyte count: > 1,500/mm3
  * Platelets: > 100,000/mm3
  * Hemoglobin: > 8.5 g/dL
  * Total bilirubin: < 1.5 mg/dL
  * Serum creatinine: < 2.5 mg/dL
  * AST or ALT: < 2.5 x institutional upper limit of normal
* Patients may have received prior radiation therapy, provided at least 4 weeks have elapsed since the conclusion of radiation therapy

Exclusion Criteria:

* Patients with biochemical only progression
* Patients who have received any prior chemotherapy for cancer of the prostate
* Patients who received antiandrogen therapy within 4 weeks prior to the first day of treatment after cessation of flutamide or nilutamide, and or within 6 weeks prior to registration after cessation of bicalutamide
* Patients receiving concomitant chemotherapy, biologic therapy, or radiation therapy
* Patients who have received Strontium 89 or other radioisotope therapies
* Patients with decreasing PSA levels following antiandrogen withdrawal
* Patients with > grade 1 peripheral sensory or motor neuropathy
* Patients with known carcinomatous meningitis or brain metastases are excluded
* Patients with past or current histories of neoplasm other than entry diagnosis except for in-situ carcinoma of any site, non-melanoma skin cancer, or other malignancy treated by surgery or radiation with a disease-free survival longer than 5 years
* Patients who have undergone major surgery < 3 weeks prior to registration, except for biopsy or placement of a venous access device. Patients must have fully recovered from all effects of any prior surgery
* Patients with histories of serious cardiac disease not adequately controlled: documented myocardial infarction within the last 6 months preceding registration, congestive heart failure, unstable angina, valvular disease with documented ventricular compromise, uncontrolled hypertension, arrhythmia uncontrolled by medication, clinically significant pericardial effusion
* Patients with active serious infections or other serious underlying medical conditions that would otherwise impair their ability to receive protocol treatments
* Patients with dementia or significantly altered mental status that would prohibit the understanding and/or giving of informed consent
* Patients receiving other investigational therapy
* Use of any investigational agent within 30 days of first day of treatment and use of Ketoconazole, hydrocortisone, glucocorticoids, or megace within 30 days of first day of treatment or other concomitant medications

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2002-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fairooz F. Kabbinavar, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of recruitment period: 10/02/2002- 5/25/2006. Types of location: Academic Medical clinics and community medical clinics. This study has 1 treatment arm; therefore randomization procedures were not utilized and all participants were enrolled to the same treatment regimen.
Groups:
- Carboplatin, Paclitaxel: Patients receive paclitaxel IV on days 1, 8, and 15 and carboplatin IV on day 1. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 4 weeks for 12 weeks and then every 2 months thereafter.
Period: Carboplatin, Paclitaxel
Arm/Group | Carboplatin, Paclitaxel
Started | 58
Completed | 45 (13 participants did not complete treatment)
Not Completed | 13
Not completed — Withdrawal by Subject | 10
Not completed — Lost to Follow-up | 1
Not completed — Death | 2
Period: Follow-up Period for Survival Status
Arm/Group | Carboplatin, Paclitaxel
Started | 45
Completed | 41
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Carboplatin, Paclitaxel
Number analyzed (Participants) | 58
Age, Continuous [Median (Full Range); unit: years] | 71 [49 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 52
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Prostate-specific Antigen (PSA) Response Rate
Description: PSA response is defined as a decline from the baseline value of >=50% confirmed by a second PSA value 4 or more weeks later.
Time Frame: Evaluated every 28 days during Treatment Period. Number of completed cycles among 58 treated patients range from 1 to 24 cycles with a median of 4.5 cycles. one cycle = 28 days.
Measure: Number; unit: participants
Arm/Group | Carboplatin, Paclitaxel
Number analyzed (Participants) | 58
participants
  Participants with PSA response | 28
  Participants with no PSA response | 30

2. Primary Outcome: Time to PSA Progression
Description: In patients whose PSA has not decreased, progressive disease is a 25% increase over the baseline value and an increase in the absolute value PSA level by >=5ng/ml, confirmed by a second value at >=4 week intervals. In patients whose PSA has decreased but has not reached response criteria, progressive disease is defined as an increase in PSA by 25% over the nadir, provided that the increase is >=5ng/ml and is confirmed by a second value at >=4 week intervals.
Time Frame: Evaluated every 28 days during Treatment Period
Measure: Median (Full Range); unit: days
Arm/Group | Carboplatin, Paclitaxel
Number analyzed (Participants) | 58
days | 115 [26 to 394]

3. Secondary Outcome: Objective Response Rate
Description: Complete response:Complete disappearance of all clinically detectable malignant disease for at least 4 weeks.Partial Response:Definite improvement in evaluable disease estimated to be in excess of 50% and agreed upon by 2 investigators. Response must last for at least 4 weeks.Stable disease:No significant change in disease for at least 4 weeks. Includes an estimated decrease of <50% and lesions with an estimated increase of <25%.Progressive disease(PD):Definite increase in area of any malignant lesion estimated to be >=25% or appearance of new lesions. Need for radiotherapy is considered PD.
Time Frame: Evaluated every 12 weeks during Treatment Period
Measure: Number; unit: participants
Arm/Group | Carboplatin, Paclitaxel
Number analyzed (Participants) | 53
participants
  Participants with Complete Response | 1
  Participants with Partial Response | 12
  Participants with Stable Disease | 33
  Participants with Progression of Disease | 7

4. Secondary Outcome: Overall Survival Rate
Description: as for outcome 3
Time Frame: Assessed every two months after completion of study treatment for 4 years
Measure: Number; unit: participants
Arm/Group | Carboplatin, Paclitaxel
Number analyzed (Participants) | 58
participants
  Deceased | 46
  Alive | 1
  Lost to Follow-up | 1
  Withdrawal by subject | 10

ADVERSE EVENTS:
Time Frame: Adverse events collected between 11/12/2002 and 08/06/2007, therefore AE reporting period is 4.7 years or 4 years and 9 months, approximately
Description: Systemic adverse event assessment occurred every 28 days through investigator assessment during treatment period and once within 30 days after last administration of study treatment.
Arm/Group | Carboplatin, Paclitaxel
Serious Adverse Events (participants affected / at risk) | 14/58
Other Adverse Events (participants affected / at risk) | 58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin, Paclitaxel (N=58)
Deep Verin Thrombosis with Pulmonary Embolism (Cardiac disorders) | 1
Paresthesia (Nervous system disorders) | 1
Subarachnoid Hemorrhage (Blood and lymphatic system disorders) | 1
Angina (Cardiac disorders) | 1
Urinary retention with acute hematuria (Renal and urinary disorders) | 1
Death secondary to cardiac arrest (Cardiac disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Anaphylaxix (Immune system disorders) | 1
Febrile Neutropenia (Infections and infestations) | 2
Hyperglycemia and diabetic management (Metabolism and nutrition disorders) | 1
Constipation (Gastrointestinal disorders) | 1
back pain (Musculoskeletal and connective tissue disorders) | 1
Gall stones (Gastrointestinal disorders) | 1
spinal injury; inability to walk or stand ultimately caused death (Nervous system disorders) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Carboplatin, Paclitaxel
Neutropenia (Blood and lymphatic system disorders) | 50/58
anemia (Blood and lymphatic system disorders) | 46/58
Alopecia (Skin and subcutaneous tissue disorders) | 45/58
Fatigue (General disorders) | 44/58
Thrombocytopenia (Blood and lymphatic system disorders) | 35/58
Neuropathy-sensory (Nervous system disorders) | 34/58
Diarrhea (Gastrointestinal disorders) | 33/58
Leukopenia (Blood and lymphatic system disorders) | 33/58
Anorexia (Gastrointestinal disorders) | 31/58
Nausea (Gastrointestinal disorders) | 30/58
Insomnia (General disorders) | 23/58
Edema, limb (Blood and lymphatic system disorders) | 22/58
constipation (Gastrointestinal disorders) | 21/58
pain, extremity-lower (General disorders) | 20/58
Pain, Not otherwise specified (General disorders) | 20/58
mood alteration-depression (Nervous system disorders) | 16/58
vomiting (Gastrointestinal disorders) | 16/58
taste alteration (Gastrointestinal disorders) | 13/58
dizziness (Nervous system disorders) | 12/58
hyperglycemia (Metabolism and nutrition disorders) | 12/58
hematuria (Renal and urinary disorders) | 11/58
hemorrhage pulmonary- nose (Blood and lymphatic system disorders) | 11/58
pain, head (General disorders) | 11/58
neuropathy-motor (Nervous system disorders) | 11/58
dyspepsia (Gastrointestinal disorders) | 9/58
fever (General disorders) | 9/58
infection-upper airway not otherwise specified (Infections and infestations) | 9/58
rash (Skin and subcutaneous tissue disorders) | 9/58
pain, back (Musculoskeletal and connective tissue disorders) | 8/58
pain, muscle (Musculoskeletal and connective tissue disorders) | 8/58
pain, shoulder (Musculoskeletal and connective tissue disorders) | 8/58
urinary frequency (Renal and urinary disorders) | 12/58
cold symptoms (General disorders) | 7/58
cough (Respiratory, thoracic and mediastinal disorders) | 7/58
infection- urinary tract not otherwise specified (Infections and infestations) | 7/58
mood alteration- anxiety (Nervous system disorders) | 7/58
allergic rhinitis (Immune system disorders) | 6/58
congestion (Respiratory, thoracic and mediastinal disorders) | 6/58
pain, abdomen (General disorders) | 6/58
sweating (General disorders) | 6/58
allergic reaction (Immune system disorders) | 5/58
ALT, elevated (Metabolism and nutrition disorders) | 5/58
dehydration (Gastrointestinal disorders) | 5/58
hypocalcemia (Metabolism and nutrition disorders) | 5/58
hypokalemia (Metabolism and nutrition disorders) | 5/58
hypotension (Cardiac disorders) | 5/58
pain, chest- non-cardiac (General disorders) | 5/58
sore throat (General disorders) | 5/58
pruritis (Skin and subcutaneous tissue disorders) | 5/58
weight loss (General disorders) | 5/58
alkaline phosphatase, elevated (Metabolism and nutrition disorders) | 4/58
AST, elevated (Metabolism and nutrition disorders) | 4/58
blurred vision (Eye disorders) | 4/58
dry mouth (Gastrointestinal disorders) | 4/58
hypoalbuminemia (Metabolism and nutrition disorders) | 4/58
Urinary retention (Renal and urinary disorders) | 4/58
cachexia (General disorders) | 3/58
pain-urination (General disorders) | 3/58
flatulence (Gastrointestinal disorders) | 3/58
flu-like syndrome (General disorders) | 3/58
gastroenteritis (Gastrointestinal disorders) | 3/58
hyperkalemia (Metabolism and nutrition disorders) | 3/58
hyperphosphatemia (Metabolism and nutrition disorders) | 3/58
hypomagnesia (Metabolism and nutrition disorders) | 3/58
hyponatremia (Metabolism and nutrition disorders) | 3/58
mucositis-oral cavity (Gastrointestinal disorders) | 3/58
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3/58
nail changes (Skin and subcutaneous tissue disorders) | 3/58
pain, bone (General disorders) | 3/58
pain, neck (General disorders) | 3/58
rigors/chills (General disorders) | 3/58
voice changes (Respiratory, thoracic and mediastinal disorders) | 3/58
dyspnea (Respiratory, thoracic and mediastinal disorders) | 12/58

LIMITATIONS AND CAVEATS:
The major weakness of the study is, it is a single-arm non-comparative study. With the small sample size of 58 participants who received treatment, the study does not have the statistical power to make categorical assessments or statements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The obligations of confidentiality shall apply for a period of 5 yrs beyond termination of Agreement between Sponsor and Investigator,but do not apply to the extent information:is or later becomes known to public;is obtained from a third party without restriction who had a legal right to disclose;is possessed by Investigators,as demonstrated by recipient's written records predating receipt from Sponsor;is required to be disclosed pursuant to a subpoena, law, regulation or other legal proceeding.